CLINICAL TRIAL: NCT06377579
Title: OBServatory of Compassionate Use of IVOsidenib in France for Patients With Acute Myeloid Leukemia
Status: Recruiting | Type: Observational
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Other Study IDs: FILObsLAM_IVOOBS
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AML in 1st line at inclusion
- AML in R/R at inclusion

SUMMARY:
Mutations in IDH genes are found in numerous cancers and more specifically in acute myeloid leukemia (AML). These mutations target specific amino acids, at positions 140 or 172 of IDH2, and 132 of IDH1. Mutant IDH proteins acquire an abnormal enzymatic activity allowing them to convert α-ketoglutarate (αKG) into D-2 hydroxyglutarate (D-2HG), an oncometabolite which massively accumulates in IDH-mutated cells. At high levels, D-2HG behaves as a competitive inhibitor of αKG and affects the activity of Fe(II)/αKG-dependent dioxygenases. This enzymatic family is involved in a broad spectrum of pathways such as demethylation of histone (JHDM histone demethylases) or DNA (methylcytosine hydroxylases of the TET family). As a result, IDH-mutated cells show altered survival, motility, invasiveness and cell differentiation. In AML, IDH1 mutations might be present in 10-15% at diagnosis

Ivosidenib (IVO) a first-in-class, oral, irreversible inhibitor of mutant IDH1 has shown clinical activity as a single agent in studies involving patients with IDH1 mutated relapsed or refractory (R/R) AML and in front line settings. In phase II clinical trials, IVO yielded 30-35% of complete response rates both in frontline and R/R settings, with long lasting responses. Based on these results, the FDA (Food and Drug Agency) gave its approval for newly-diagnosed AML IDH1mut patients who are ≥ 75 years old or who have comorbidities and in R/R. However, European Medicines Agency (EMA)'s did not approved IVO due to lack of evidences to support the application. Agios Netherlands B.V. (the company that previously own the drug before Servier Laboratories) withdrew its EMA application. Nevertheless, IVO has been available in France through a compassionate use program (CUP), since February 2020 for R/R patients and March 2022 for first line treatment.

In this multicentric retrospective study, sponsor aim to evaluate the efficacy and safety of Ivo in two cohorts of IDH1mut AML patients treated within the CUP. The first cohort will concern patients treated in first line setting and the second cohort those treated in R/R disease. Results might provide new insights regarding IVO in real life settings and support signs of efficacy. This could provide new data for the haematologist community and for another appliance to grant EMA approval of IVO in the setting of R/R IDH1mut AML.

ELIGIBILITY:
Inclusion Criteria:

* Patient with IDH1 R132 mutated with newly diagnosed or Relapsed or Refractory (R/R) acute myeloid leukemia
* Patient treated within French compassionate access program that have started the treatment between 01/01/2017 to 01/08/2023
* patient treated by Ivosidenib received either as a monotherapy or in combination with other AML therapy (i.e. azacytidine, venetoclax)
* Patient not included within IDH inhibitor clinical trial.

Exclusion Criteria:

* Patients who expressed their opposition to entered in the study
* Patients who received IVO through a trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years old or more, with newly diagnosed or relapsed or refractory IDH1 mutated AML according to ELN 2022 and treated with IVO thanks to the CUP between the period 01/01/2017 to 01/08/2023, treated in French AML FILO or ALFA centers
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
characterize the Overall survival (OS) in the both cohort : 1st line and Relapsed/Refractory (R/R) | 6 months
  defined as the time from date of initiation of Ivosidebib to date of death due to any cause.
  Patients still alive or lost to follow up will be censored at the time they were last known to be alive

SECONDARY OUTCOMES:
characterize the composite response rate (CRc) at any time during follow-up, for the both cohort : 1st line and Relapsed/Refractory (R/R) | 6 months
  CRc is defined as the sum of Complete remission (CR) + Complete remission with partial hematological recovery (CRh) + Complete remission with incomplete count recovery (CRi) + MLFS, according to ELN 2022 criteria
characterize the Event Free Survival (EFS) in both cohorts : 1st line and Relapsed/Refractory (R/R) | 6 months
  defined as the time from initiation of Ivosidenib (IVO) to the date of treatment failure, hematologic relapse from Complete remission (CR)/Complete remission with partial hematological recovery (CRh)/ Complete remission with incomplete count recovery (CRi)/ Morphologic leukemia-free state (MLFS) or death from any cause, whichever occurs first; Treatment failure is defined as not achieving either CR, CRh,CRi or MLFS by day 180 from Ivo start
characterize the incidence and relatedness of serious adverse events (SAE), for patients treated by Ivosidenib, for both cohorts : 1st line and Relapsed/Refractory (R/R) | 6 months
  description of grade 3/4 SAE and death according to CTCAE v5
describe the management of treatment by Ivosidenib in both cohorts : 1st line and Relapsed/Refractory (R/R) | 6 months
  daily dose of Ivosidenib, description of Ivosidenib dose modification
describe the management of treatment by Ivosidenib in both cohorts : 1st line and Relapsed/Refractory (R/R) | 6 months
  duration of treatment by Ivosidenib

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PETERLIN, Dr, Principal Investigator — French Innovative Leukemia Organisation
Locations (21):
- France (21):
  - Amiens CHU, Amiens
  - Angers CHU, Angers
  - Bayonne CH, Bayonne
  - Besançon CHU, Besançon
  - CHU Estaing, Clermont-Ferrand
  - Créteil CHU HENRI MONDOR, Créteil
  - DUNKERQUE-Hôpital Alexandra Lepève, Dunkirk
  - Grenoble CHU, Grenoble
  - Le Mans CH, Le Mans
  - Lyon sud CHU, Lyon
  - Marseille IPC, Marseille
  - Meaux CH de l'Est francilien, Meaux
  - Montpellier - Chu Saint Eloi, Montpellier
  - Mulhouse Chu, Mulhouse
  - Nantes CHU, Nantes
  - Nice CHU, Nice
  - Orléans CHU, Orléans
  - Paris Saint Louis, Paris
  - Bordeaux CHU, Pessac
  - ICANS - Institut de cancérologie de strasbourg europe, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse

IPD SHARING:
Plan to Share IPD: No